CLINICAL TRIAL: NCT06557538
Title: Comparing the Ankle Brachial Pressure Index Score of Automatic ABPI Device vs Manual ABPI Device to Classify Lower Limb Ulcers and Guide Treatment in Patients Under Community Services
Brief Title: A Comparison of Automatic ABPI vs Manual ABPI Device Scores
Status: Active, not recruiting | Type: Observational
Sponsor: University of Southampton (Other)
Collaborators: Berkshire Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ERGO 92967
Record Dates: First submitted 2024-08-07; First posted 2024-08-16 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-09

CONDITIONS: Lower Limb Ulcers
Keywords: Lower limb ulcers; Automatic ankle brachial pressure index; MESI MD ABPI; Huntleigh dopplex; Community; Comparison; ABPI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- People over the age of 18 with lower limb ulcers under Community Services: Comparison of reading between automatic and manual device ABPI scores
  Interventions: Device: Automatic Ankle Brachial Pressure Index device assessment; Device: Manual Ankle Brachial Pressure Index assessment

INTERVENTIONS:
Device: Automatic Ankle Brachial Pressure Index device assessment — The automatic device assesses 3 limbs, providing automatic simultaneous ABPI measurement of systolic, diastolic and mean arterial blood pressure on to calculate the patient's ABPI (Medi UK 2022).
Device: Manual Ankle Brachial Pressure Index assessment — The manual device assesses 4 limbs, providing brachial, ankle and pedal systolic pressures. A simple calculation is then made by the clinician to determine the ratio of ankle and brachial systolic pressure (ABPI) (Day 2015).

SUMMARY:
The aim of the study is to compare the Ankle Brachial Pressure Index (ABPI) scores of two devices. The two devices that will be compared are the MESI MD ABPI automatic device and the Huntleigh Dopplex manual device.

The Huntleigh Dopplex manual device is widely used, though the MESI MD ABPI automatic devices can reduce waiting times, reduce discomfort for patients and save nursing time. ABPI devices provide a score that supports nurses to provide suitable treatment for patients with a lower limb ulcer.

In the community, patients with lower limb ulcers are offered an ABPI assessment and then treatment is decided based on the score. Participants will be patients with lower limb ulcers referred to community nursing for a lower limb and ABPI assessment. At their routine appointment patients will have a manual assessment and an automatic assessment, and the results will be compared. The study will take place in the county of Berkshire either in patients' homes or in the lower limb clinic. Registered nurses will undertake all assessments. The direct care part of the study will run from July 2024 - December 2024. The data will be pseudonymised, and the findings written as a report that may be sent for publishing.

DETAILED DESCRIPTION:
A lower limb ulcer is defined as a non-healing wound, venous disease being the most common cause and the gold standard treatment is compression therapy. The estimated cost implication of managing wounds in the UK is more than £5 billion per year with much of that cost coming from Nursing time and resources Wounds UK classify lower limb ulcers as either a 'Simple venous lower limb ulcer' or 'Complex venous ulcer'. National Institute for Health and Care Excellence states that lower limb ulcer assessments should be holistic including, lower limb, and wound assessments to enable early intervention, increase healing rates, and reduce financial burden. Patients should have an Ankle Brachial Pressure Index (ABPI) measurement assessment which will then give a clinical result to support classification of lower limb ulcers and to establish whether compression therapy is appropriate.

Historically, ABPI has been measured manually using a handheld doppler. This method can be time consuming, unreliable and requires a skilled clinician to undertake it. The test takes between 30 minutes to 1 hour and can also cause significant discomfort for patients with lower limb ulcers as cuffs are placed on limbs and inflated up to four times on each.

With the increasing cost and ageing population, it has been identified that healthcare professionals should be aware of advances in technology and use devices available that are more efficient, providing better patient outcomes. With that said, new automated devices have become available and have been used in community trusts since November 2022. These devices are more time efficient, user friendly and more comfortable for people with lower limb ulcers. The MESI MD ABPI device was introduced into Berkshire Healthcare NHS Foundation Trust (BHFT) in November 2022.

In 2022 NHS England (NHSE) published a Commissioning for Quality and Innovation (CQUIN) guidance with CQUIN targets aimed at ensuring robust, quality wound assessment and reducing deficiencies in intervention and care for patients with lower limb ulcers.

The NHSE CQUIN require 50% of patients with lower limb wound(s) to have a full clinical assessment within 28 days of initial wound presentation and have compression therapy of 40mmHg applied. Following the introduction of the MESI MD ABPI automatic devices to BHFT, the CQUIN achievement results increased by 10%.

Due to the impact of introducing the MESI MD ABPI device BHFT wished to continue with their use. NICE published the guidance on usage of automatic ABPI measurement devices in people with lower limb ulcers. They identified that there is a lack of evidence on the accuracy of automated ABPI devices. They provided a criterion for Trusts who want to continue using these devices. It was identified that the trust met all NICE criteria except for Criteria. Therefore, BHFT agreed to support an research study project on the MESI MD ABPI device to compare its agreement with results of the manual doppler.

As an advanced clinician expected to be competent in the four pillars of advanced practice including research, I agreed this would be an appropriate study for me to undertake as it would benefit both my development, and patients under our care.

NICE Criterion for continued use of automatic ABPI devices.

1. People using the devices have experience assessing peripheral arterial disease.
2. People using the devices are aware of their limitations, particularly diagnostic accuracy, and the risk of missing peripheral arterial disease, and that there are differences between devices.
3. Further assessment using other methods, including manual doppler, is available.
4. Trusts using devices collect data or do research to assess their value and how well they identify people with peripheral arterial disease.

NICE advised that future research on automated ABPI devices should:

1. Assess their ability to detect peripheral arterial disease in people with leg ulcers
2. Assess how they affect time to treatment for venous leg ulcers
3. Assess clinical outcomes for treatments started after ABPI assessment
4. Explore the most appropriate user (specialist and non-specialist in assessing peripheral arterial disease) and the most appropriate healthcare setting for their use
5. Explore whether different ABPI thresholds can improve their sensitivity for detecting peripheral arterial disease.

There are several studies and anecdotal evidence that the automatic devices save time and reduce time to treatment in line with CQUIN standards. However, there is dearth of research on the efficacy of the automatic devices and therefore, it was decided to undertake a study on comparing the results of the automatic to the validated manual device to fulfil criteria one.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years old
* Participants will have at least one lower limb ulcer
* Participants will have capacity to consent
* Participants will live in the Geographical area of Berkshire

Exclusion Criteria:

* Participants found on assessment to have monophasic pulse sounds or signs of aortic stenosis
* Patients deemed to not have capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with an open referral to Berkshire community services, living in the county of Berkshire with a lower limb ulcer.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Ankle Brachial Pressure score | Through study completion of average of 7 months
  Difference between ABPI scores from automatic and manual ABPI device.

SECONDARY OUTCOMES:
Difference in lower limb ulcer classification | Through study completion of average of 7 months
  Difference in lower limb ulcer classification between automatic and manual ABPI device.

CONTACTS AND LOCATIONS:
Overall Officials: Jamal Hossain, PHD, Study Chair — School of Health Sciences,University of Southampton,Highfield Campus,University Road,Soton SO17 1BJ
Locations (1):
- Berkshire Healthcare NHS Foundation Trust, Bracknell, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be held in the University repository and be available for use in future study.
Supporting Information: SAP, CSR, Analytic Code
Time Frame: Anonymous data indefinitely
Access Criteria: Researchers connected with the University of Southampton and Berkshire Healthcare Foundation Trust.
URL: https://www.southampton.ac.uk/research/researcher-support.page

REFERENCES:
- [Background] Al-Qaisi M, Nott DM, King DH, Kaddoura S. Ankle brachial pressure index (ABPI): An update for practitioners. Vasc Health Risk Manag. 2009;5:833-41. doi: 10.2147/vhrm.s6759. Epub 2009 Oct 12. PMID 19851521
- [Background] Boast, G., Green, J., Chambers, R. and Calderwood, R. (2019) 'Improving assessment and management of lower limb wounds', Journal of community nursing,33 (5), pp. 34 - 38
- [Background] Benbow M. An introduction and guide to effective Doppler assessment. Br J Community Nurs. 2014 Dec;Suppl Wound Care:S21-6. doi: 10.12968/bjcn.2014.19.Sup3.S21. PMID 25478852
- [Background] Buxey, K. (2020) 'Introducing MESI ABPI MD automated device to a leg club setting', Journal of Community Nursing, 34 (1), pp. 22- 26
- [Background] Day J. Diagnosing and managing venous leg ulcers in patients in the community. Br J Community Nurs. 2015 Dec;20 Suppl 12:S22-30. doi: 10.12968/bjcn.2015.20.Sup12.S22. PMID 26639070
- [Background] Dowsett, C. and Taylor, C. (2018) 'Reducing variation in leg ulcer assessment management using quality improvement methods', Wounds UK, 14 (4), pp. 46 - 51
- [Background] Boyers, D., Cruickshank, M., Aucott, L., Kennedy, C., Manson, P., Bachoo, P. and Brazelli, M (2022) Automated measurement of ankle brachial pressure index for assessing the presence of peripheral arterial disease in people with leg ulceration, University of Aberdeen Report. Available at: diagnostics-assessment-report
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Grove, SK., Gray, JR. and Burns, N. (2019) Understanding Nursing Research: Building an Evidence-Based Practice. St. Louis, Missouri: Elsevier
- [Background] Lloyd- Jones, M. (2019) 'Wound Care: What's new? 1. Ankle and brachial pressure index in practice', British journal of Healthcare Assistants, 13 (9), pp. 422- 426
- [Background] Medi UK Ltd. (2022) Instructions for use: MESI ABPI MD, Ankle Brachial Pressure Index. Available at: www.mediuk.co.uk
- [Background] Moffat, C., Martin, R. and Smithdale, R. (2007) Leg Ulcer Management. Oxford: Blackwell publishing
- [Background] National Health Service England (NHSE) (2022) Commissioning for Quality and Innovation (CQUIN): 2023/24 guidance. Available at: https://www.england.nhs.uk/nhs-standard-contract/cquin/cquin-23-24/
- [Background] Guest JF, Ayoub N, McIlwraith T, Uchegbu I, Gerrish A, Weidlich D, Vowden K, Vowden P. Health economic burden that wounds impose on the National Health Service in the UK. BMJ Open. 2015 Dec 7;5(12):e009283. doi: 10.1136/bmjopen-2015-009283. PMID 26644123
- [Background] Lindsay, E. and Whiteley, M. (2018) A partnership approach: helping patients with leg ulcers and varicose veins', Wounds UK, 14 (3), pp. 86- 88
- [Background] Rayaa, R., Martíneza, N., Cayuelasa, F., Perab, G. and García, Y. (2019) 'Comparison of two automatic oscillometers vs the traditional method with Doppler probe in the determination of the ankle brachial index', Atencion Primaria Practica, 1(1), pp 3- 8
- [Background] Span M, Gersak G, Millasseau SC, Meza M, Kosir A. Detection of peripheral arterial disease with an improved automated device: comparison of a new oscillometric device and the standard Doppler method. Vasc Health Risk Manag. 2016 Jul 29;12:305-11. doi: 10.2147/VHRM.S106534. eCollection 2016. PMID 27536125
- [Background] Wounds UK (2016) Best Practice Statement: Holistic Management of Venous Leg Ulceration. Available at: Venous Leg Ulceration.indd (wounds-uk.com)
- [Background] University of Southampton (2012) University Ethics Policy. Available at: University Ethics Policy | University of Southampton
- [Background] Wounds UK (2019) Best Practice Statement Ankle Brachial pressure index (ABPI) in practice. Available at https://wounds-uk.com/best-practice-statements/ankle-brachial-pressure-index-abpi-practice/
- See also: NICE guidance relevant to study background — https://www.nice.org.uk/guidance/cg147
- See also: NICE guidance relevant to study background — https://www.nice.org.uk/guidance/dg52
- See also: CQUIN guidance — http://www.england.nhs.uk/nhs-standard-contract/cquin/cquin-23-24/